CLINICAL TRIAL: NCT05501821
Title: A Phase I, First-in-human, Multicenter, Open-label, Dose Escalation Followed by an Expansion Phase Clinical Study of KBA1412 Given as Monotherapy or in Combination With Pembrolizumab in Adults With Advanced Solid Malignant Tumors
Brief Title: Study of KBA1412 in Participants With Advanced Solid Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kling Biotherapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KBA1412-101
Record Dates: First submitted 2022-08-04; First posted 2022-08-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor Malignancy
Keywords: solid tumor adult; refractory cancer
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Part A will consist of multiple cohorts, each at an escalated dose level of KBA1412.
  Part B will consist of disease specific cohorts, each cohort treated with KBA1412 at a fixed dose level.
  Part C will consist of disease specific cohorts, each cohort treated with KBA1412 at a fixed dose in combination with pembrolizumab at a fixed dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A, dose escalation monotherapy (Experimental): KBA1412 monotherapy, given intravenously, Q3W, multiple dose levels
  Interventions: Drug: KBA1412
- Part B, expansion monotherapy (Experimental): KBA1412 monotherapy, given intravenously, Q3W, at fixed dose as defined in dose-escalation phase (Part A)
  Interventions: Drug: KBA1412
- Part C, expansion combination therapy (Experimental): KBA1412 in combination with pembrolizumab, given intravenously, Q3W, KBA1412 at fixed dose as defined in dose-escalation phase (Part A), Pembrolizumab at fixed dose
  Interventions: Drug: KBA1412; Drug: Pembrolizumab

INTERVENTIONS:
Drug: KBA1412 — Part A, B, C
Drug: Pembrolizumab — Part C only
  Other Names: Keytruda
  Arms: Part C, expansion combination therapy

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of KBA1412, a patient derived, fully human, monoclonal antibody targeting CD9, in patients with advanced solid malignant tumors

DETAILED DESCRIPTION:
Patient interested in participation in a clinical study will be informed about the study and potential risks, all patients giving written informed consent will undergo a 3-week screening period to determine their eligibility for entry in the study. Patients will receive KBA1412 or KBA1412 in combination with pembrolizumab.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients aged ≥18 years.
* Histologically and/or cytologically confirmed locally advanced or metastatic solid tumors refractory to standard therapy or for whom no standard therapy is available.
* For Parts B and C, patients for whom anti-PD-1 or anti-programmed cell death ligand 1 (anti-PD-L1) are the SOC should have progressed on these therapies before being eligible for enrollment in Parts B and C. Patients cannot have received more than one anti-PD-1 or anti-PD-L1 based regimen.
* Disease accessible for core needle biopsy both pre- and post-treatment with KBA1412. Biopsies will be mandatory for patients with melanoma and required for other tumor types depending on feasibility of obtaining tissue.
* Measurable disease defined as: At least 1 lesion of ≥10 mm in the longest diameter for a non lymph node or ≥15 mm in the short-axis diameter for a lymph node that is serially measurable according to iRECIST using CT/MRI and will not be used for on-study paired biopsies.
* ECOG Performance Status of 0-1.
* Adequate hematologic, renal and hepatic function

Exclusion criteria:

* History of severe hypersensitivity reactions to other monoclonal antibodies.
* Prior treatment with:

  * Any chemotherapy, anticancer small molecule therapy or investigational drug or device within 14 days or 5 half-lives (whichever is longer) prior to study treatment administration
  * Biological agents (including monoclonal antibodies) within 28 days prior to study treatment administration
  * Radiation, within 14 days prior to study treatment administration
  * Treatment with nitrosoureas or mitomycin C require a 42-day washout prior to study treatment administration
  * Anti-CD40 antibody or with FMS-like tyrosine kinase 3 ligand (FLT3L)
  * KBA1412.
* Major surgery or significant traumatic injury within 4 weeks prior to study treatment administration.
* Excluding the primary tumor leading to enrollment in this study, any other active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the bladder or cervix) within 24 months prior to study treatment administration.
* Untreated primary central nervous system (CNS) malignancy.
* Use of immunosuppressive medications within 4 weeks or systemic corticosteroids at doses exceeding 10 mg/ day (prednisone equivalent) within 2 weeks prior to study treatment administration.
* Active autoimmune disease that has required systemic treatment within 2 years prior to study treatment administration.
* Clinically significant cardiovascular disease, e.g., cerebral vascular accident/stroke or myocardial infarction, within 6 months prior to study treatment administration, unstable angina, congestive heart failure (New York Heart Association [NYHA] Class ≥III), or unstable cardiac arrhythmia requiring medication.
* History of a major bleeding event (requiring a blood transfusion of >2 units) not related to a tumor within 12 months prior to study treatment administration.
* Ongoing Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 toxicity related to a previously administered anticancer agent with the following exceptions:

  * CTCAE Grade 2 neuropathy or alopecia
  * CTCAE Grade 2 immune-related endocrinopathy attributed to a checkpoint inhibitor and controlled with hormone replacement alone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Part A & B & C: Frequency and severity of AEs as assessed by CTCAE v5.0 | Through study completion, an average of 1 year
  Monitoring incidence and severity of Adverse Events during trial participation for each participant
Part A: Frequency and type of DLT s using the CTCAE v5.0 | First 21 days of treatment
  A DLT is defined as an adverse event that is unrelated to disease progression, intercurrent illness, or concomitant medications and is occurring during the first 21 days of treatment. These events will be classified according to the CTCAE v5.0
Number of participants with an antitumor response to KBA1412 monotherapy (Part B) or to KBA1412 in combination with pembrolizumab (Part C) | Approximately 24 weeks
  Response according to immune Response Evaluation Criteria in Solid Tumors (iRECIST)

SECONDARY OUTCOMES:
Part A: Number of participants with an antitumor response to KBA1412 monotherapy | Approximately 24 weeks
  Response according to immune Response Evaluation Criteria in Solid Tumors (iRECIST)
Pharmacokinetic of KBA1412 monotherapy (Part A & B) and KBA1412 in combination with pembrolizumab (Part C), area under the concentration versus time curve (AUC) | Approximately 24 weeks
  Area under the plasma concentration versus time curve (AUC) of KBA1412 will be assessed in all participants
Incidence and prevalence of anti-KBA1412 antibodies for KBA1412 monotherapy (Part A & B) and KBA1412 in combination with pembrolizumab (Part C) | Approximately 24 weeks
  Development of antibodies (anti-drug antibodies) to KBA1412 will be evaluated for all participants
Change in biomarkers for KBA1412 monotherapy (Part A & B) and KBA1412 in combination with pembrolizumab (Part C) pre- and post-dose in tumor tissue | Approximately 24 weeks
  Change in pharmacodynamic properties of KBA1412 pre- and post-dose in immune infiltration, activation and cytotoxicity assessed by Immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - University Hospital Ghent, Ghent
- Netherlands (3):
  - Dutch Cancer Institute AVL, Amsterdam
  - University Hospital Leiden (LUMC), Leiden
  - Erasmus Medical Center Rotterdam, Rotterdam

IPD SHARING:
Plan to Share IPD: No